CLINICAL TRIAL: NCT00004323
Title: Phase II Study of Bone Marrow Transplantation Using Related Donors in Patients With Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of California, Los Angeles (Other)
Purpose: Treatment
Other Study IDs: 199/11863; UCLA-94020602
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-04

CONDITIONS: Aplastic Anemia
Keywords: aplastic anemia; hematologic disorders; rare disease
MeSH Terms: conditions — Anemia, Aplastic; Hematologic Diseases; Rare Diseases | interventions — Antilymphocyte Serum; Cyclophosphamide; Cyclosporine; Mesna; Methotrexate; Methylprednisolone

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: cyclophosphamide
Drug: cyclosporine
Drug: mesna
Drug: methotrexate
Drug: methylprednisolone

SUMMARY:
OBJECTIVES: I. Evaluate the efficacy of related, HLA-identical bone marrow transplantation following cyclophosphamide (CTX) and antithymocyte globulin in patients with aplastic anemia.

II. Evaluate the efficacy of related, HLA-nonidentical bone marrow transplantation following CTX and total-body irradiation/total-lymphoid irradiation in patients with aplastic anemia.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients with HLA-identical donors receive cyclophosphamide/mesna, antithymocyte globulin (ATG), and methylprednisolone (MePRDL), followed by allogeneic marrow transplantation.

Patients with HLA-nonidentical (5/6 or 4/6) donors and those with a systemic reaction to ATG receive the same dosage of myeloablative chemotherapy and rescue. In addition, these patients are treated with total-body irradiation, total-lymphoid irradiation, and methotrexate.

All patients received MePRDL and cyclosporine for graft-versus-host prophylaxis.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Severe aplastic anemia with 2 of the following criteria: Polymorphonuclear neutrophils no more than 0.5 x 10 to the ninth/L Platelets no more than 20 x 10 to the ninth/L Reticulocytes no more than 30 x 10 to the ninth/L Hypocellular bone marrow Related donor aged 6 weeks or more, matching at least 4 of 6 HLA A, B, and DRI loci, as follows: HLA-identical family member for patients aged less than 40 years HLA-nonidentical family member for patients aged less than 55 years failing antithymocyte globulin or other immunosuppressive therapy The following eligible for transplantation as initial therapy: Patients aged less than 40 years with HLA-matched donor Patients aged 40-45 years with HLA-identical donor No neoplastic or preneoplastic evolution --Patient Characteristics-- Age: Under 40 (55 if ATG failure) Hepatic: No severe liver dysfunction Renal: No severe renal dysfunction Cardiovascular: No severe cardiac dysfunction Other: No other organ dysfunction that would compromise survival after transplant No HIV infection

Ages: 0 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10
Dates: Start 1995-02

CONTACTS AND LOCATIONS:
Overall Officials: Mary Carol Territo, Study Chair — University of California, Los Angeles
Locations (1):
- Center for Health Sciences, Los Angeles, California, United States